CLINICAL TRIAL: NCT06360523
Title: ProstateAI - A Prospective Paired Validating Cohort Study to Evaluate an MRI-based Optimized Prostate Cancer Diagnostic Pathway Powered by Artificial Intelligence
Brief Title: To Evaluate an MRI-based Optimized Prostate Cancer Diagnostic Pathway Powered by Artificial Intelligence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Associate Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CRE-2024.141
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: AI review (index) and radiologist review (standard) will be blinded to each other, while biopsy urologists will be well-informed of the findings of both AI review and radiologist review and make personalized biopsy plan by combining both findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI review (index) (Experimental): self-paired design, AI review (index)
  Interventions: Diagnostic Test: AI modal
- Radiologist review (Standard) (Active Comparator): self-paired design, radiologist review (standard)
  Interventions: Diagnostic Test: Standard review

INTERVENTIONS:
Diagnostic Test: AI modal — The MRI image will be reviewed by radiologist and AI model(s) respectively. The urologist will combine the results of the two approaches to optimize the biopsy strategy which is expected to result in more accurate diagnosis.
  Arms: AI review (index)
Diagnostic Test: Standard review — The MRI image will be reviewed by radiologist.
  Arms: Radiologist review (Standard)

SUMMARY:
It is a prospective paired-cohort study for diagnostic test evaluation. The study aim to determine the accuracy of AI review and investigate whether AI review could detect MRI visible significant cancer as effective as radiologist review. MRI image of about 368 men recommended for biopsy will be reviewed by an AI model and an experienced radiologist, respectively. AI review (index) and radiologist review (standard) will be blinded to each other, while biopsy urologists will be well-informed of the findings of both AI review and radiologist review and make personalized biopsy plan by combining both findings. The pathological results of MRI-ultrasound fusion biopsy (reference) will serve as the gold standard to assess the diagnostic accuracy.

DETAILED DESCRIPTION:
ProstateAI is a prospective paired-cohort study for diagnostic test evaluation. ProstateAI will determine the accuracy of AI review and investigate whether AI review could detect MRI visible significant cancer as effective as radiologist review. MRI image of about 368 men recommended for biopsy will be reviewed by an AI model and an experienced radiologist, respectively. AI review (index) and radiologist review (standard) will be blinded to each other, while biopsy urologists will be well-informed of the findings of both AI review and radiologist review and make personalized biopsy plan by combining both findings. The pathological results of MRI-ultrasound fusion biopsy (reference) will serve as the gold standard to assess the diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients recommended for prostate biopsy for diagnosis or re-assessment.
* Men at least 18 years or over
* Patients with prostate MRI image eligible for radiologist review and AI review.
* Patient Informed Consent is signed.

Exclusion Criteria:

* Patient contraindicated to prostate biopsy
* Patient failed to complete the biopsy procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 368 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Prostate Cancer detection rate of ISUP grade group ≥2 | Through study completion, an average of 1 year
  Assessed by AI review, Radiologist review, and Biopsy (Targeted).

SECONDARY OUTCOMES:
Diagnosis of any grade of prostate cancer | Through study completion, an average of 1 year
  Assessed by prostate biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Peter CHIU, FRCS, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halabi S, Lin CY, Kelly WK, Fizazi KS, Moul JW, Kaplan EB, Morris MJ, Small EJ. Updated prognostic model for predicting overall survival in first-line chemotherapy for patients with metastatic castration-resistant prostate cancer. J Clin Oncol. 2014 Mar 1;32(7):671-7. doi: 10.1200/JCO.2013.52.3696. Epub 2014 Jan 21. PMID 24449231
- [Background] Ilic D, Djulbegovic M, Jung JH, Hwang EC, Zhou Q, Cleves A, Agoritsas T, Dahm P. Prostate cancer screening with prostate-specific antigen (PSA) test: a systematic review and meta-analysis. BMJ. 2018 Sep 5;362:k3519. doi: 10.1136/bmj.k3519. PMID 30185521
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Background] Wei JT, Barocas D, Carlsson S, Coakley F, Eggener S, Etzioni R, Fine SW, Han M, Kim SK, Kirkby E, Konety BR, Miner M, Moses K, Nissenberg MG, Pinto PA, Salami SS, Souter L, Thompson IM, Lin DW. Early Detection of Prostate Cancer: AUA/SUO Guideline Part II: Considerations for a Prostate Biopsy. J Urol. 2023 Jul;210(1):54-63. doi: 10.1097/JU.0000000000003492. Epub 2023 Apr 25. PMID 37096575
- [Background] Bass EJ, Pantovic A, Connor MJ, Loeb S, Rastinehad AR, Winkler M, Gabe R, Ahmed HU. Diagnostic accuracy of magnetic resonance imaging targeted biopsy techniques compared to transrectal ultrasound guided biopsy of the prostate: a systematic review and meta-analysis. Prostate Cancer Prostatic Dis. 2022 Feb;25(2):174-179. doi: 10.1038/s41391-021-00449-7. Epub 2021 Sep 21. PMID 34548624
- [Background] Siddiqui MM, Rais-Bahrami S, Truong H, Stamatakis L, Vourganti S, Nix J, Hoang AN, Walton-Diaz A, Shuch B, Weintraub M, Kruecker J, Amalou H, Turkbey B, Merino MJ, Choyke PL, Wood BJ, Pinto PA. Magnetic resonance imaging/ultrasound-fusion biopsy significantly upgrades prostate cancer versus systematic 12-core transrectal ultrasound biopsy. Eur Urol. 2013 Nov;64(5):713-719. doi: 10.1016/j.eururo.2013.05.059. Epub 2013 Jun 12. PMID 23787357
- [Background] Wegelin O, van Melick HHE, Hooft L, Bosch JLHR, Reitsma HB, Barentsz JO, Somford DM. Comparing Three Different Techniques for Magnetic Resonance Imaging-targeted Prostate Biopsies: A Systematic Review of In-bore versus Magnetic Resonance Imaging-transrectal Ultrasound fusion versus Cognitive Registration. Is There a Preferred Technique? Eur Urol. 2017 Apr;71(4):517-531. doi: 10.1016/j.eururo.2016.07.041. Epub 2016 Aug 25. PMID 27568655
- [Background] Wei C, Szewczyk-Bieda M, Bates AS, Donnan PT, Rauchhaus P, Gandy S, Ragupathy SKA, Singh P, Coll K, Serhan J, Wilson J, Nabi G. Multicenter Randomized Trial Assessing MRI and Image-guided Biopsy for Suspected Prostate Cancer: The MULTIPROS Study. Radiology. 2023 Jul;308(1):e221428. doi: 10.1148/radiol.221428. PMID 37489992
- [Background] Annamalai A, Fustok JN, Beltran-Perez J, Rashad AT, Krane LS, Triche BL. Interobserver Agreement and Accuracy in Interpreting mpMRI of the Prostate: a Systematic Review. Curr Urol Rep. 2022 Jan;23(1):1-10. doi: 10.1007/s11934-022-01084-y. Epub 2022 Feb 28. PMID 35226257
- [Background] Schergna E, Armani M. [Muscular diseases: epidemiology of progressive muscular dystrophies]. Minerva Med. 1981 Apr 28;72(17):1045-9. Italian. PMID 6939970
- [Background] Lenfant L, Beitone C, Troccaz J, Roupret M, Seisen T, Voros S, Mozer PC. Learning curve for fusion magnetic resonance imaging targeted prostate biopsy and three-dimensional transrectal ultrasonography segmentation. BJU Int. 2024 Jun;133(6):709-716. doi: 10.1111/bju.16287. Epub 2024 Jan 31. PMID 38294145
- [Background] Halstuch D, Baniel J, Lifshitz D, Sela S, Ber Y, Margel D. Characterizing the learning curve of MRI-US fusion prostate biopsies. Prostate Cancer Prostatic Dis. 2019 Dec;22(4):546-551. doi: 10.1038/s41391-019-0137-2. Epub 2019 Mar 6. PMID 30842585
- [Background] Kasabwala K, Patel N, Cricco-Lizza E, Shimpi AA, Weng S, Buchmann RM, Motanagh S, Wu Y, Banerjee S, Khani F, Margolis DJ, Robinson BD, Hu JC. The Learning Curve for Magnetic Resonance Imaging/Ultrasound Fusion-guided Prostate Biopsy. Eur Urol Oncol. 2019 Mar;2(2):135-140. doi: 10.1016/j.euo.2018.07.005. Epub 2018 Aug 17. PMID 31017088
- [Background] Bhattacharya I, Khandwala YS, Vesal S, Shao W, Yang Q, Soerensen SJC, Fan RE, Ghanouni P, Kunder CA, Brooks JD, Hu Y, Rusu M, Sonn GA. A review of artificial intelligence in prostate cancer detection on imaging. Ther Adv Urol. 2022 Oct 10;14:17562872221128791. doi: 10.1177/17562872221128791. eCollection 2022 Jan-Dec. PMID 36249889
- [Background] Lomas DJ, Ahmed HU. All change in the prostate cancer diagnostic pathway. Nat Rev Clin Oncol. 2020 Jun;17(6):372-381. doi: 10.1038/s41571-020-0332-z. Epub 2020 Feb 28. PMID 32112055